CLINICAL TRIAL: NCT05154877
Title: Evaluation of the Quality of Images and the Sensitivity of Detection of Sub-Centimeter Lesions of a New Generation of PET-CT OMNI
Brief Title: Evaluation of a New Generation of PET-CT OMNI
Status: Completed | Type: Observational
Sponsor: GE Healthcare (Industry)
Collaborators: Institut Claudius Regaud (Other)
Responsible Party: Sponsor
Other Study IDs: 209658964
Record Dates: First submitted 2021-11-01; First posted 2021-12-13 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Oncology
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- DMI5R: The subject will undergo two PET/CT scans: one on the DMI5R scanner and one on the OMNI scanner.
  Interventions: Device: OMNI PET/CT Scan
- DIQ5R: The subject will undergo two PET/CT scans: one on the DIQ5R scanner and one on the OMNI scanner.
  Interventions: Device: OMNI PET/CT Scan

INTERVENTIONS:
Device: OMNI PET/CT Scan — The subject will undergo two PET/CT scans: one on the standard of care scanner and one on the OMNI scanner.

SUMMARY:
The overarching purpose of the study is to provide supporting evidence to the value proposition of OMNI, that offers global access to an affordable hybrid PET/CT system similar in performance to that of systems utilized by world-class academic centers. Specifically, the study will collect a library of oncology 18FDG PET image data from the OMNI system and evaluate the images as compared to the standard of care PET/CT systems.

This evaluation is being performed as a necessary part of product development in order to obtain user feedback on device performance, user preference, image quality (IQ), workflow, and new device features. This study will also help to inform protocol development in reducing both scan time and radiologic tracer dose.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old;
2. A clinical indication for Fluorodeoxyglucose (FDG or 18F-FDG) PET/CT examination according to current clinical practice standards;
3. Have ≥ 1 WHO Karnofsky index < 70;
4. Are able to maintain a supine position twice;
5. Are affiliated with a Social Security scheme in France; AND,
6. Are able and willing to provide informed consent for participation in this study, per the EC approved policy.

Exclusion Criteria:

1. Have uncontrolled diabetes;
2. Have a formal contraindication to certain imaging examinations (i.e., significant claustrophobia, or other contraindications as determined by the ordering physician.)
3. Are known to be pregnant or breastfeeding (the investigational site will follow their standard practice of verifying for women of childbearing age; OR,
4. Are known to have any psychological, family, geographic, or sociological condition that does not allow compliance with the medical monitoring and/or the procedures provided for in the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects having an indication for FDG or 18F-FDG PET/CT examination according to current clinical practice standards will be enrolled in this study. These subjects are representative of the general population that is expected to use the device in clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2022-05-30 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2023-12-18 (Actual)

PRIMARY OUTCOMES:
Evaluation | through study completion, an average of 1 year
  Completed image evaluation will be completed using a 5 point Likert Scale of the OMNI system in comparison to the SoC systems for the same subjects, including analysis, reading, and scoring utilizing Likert Scaling and preference questions by three (3) qualified Nuclear Medicine Physicians. Likert scale is 1-5, 3,4 & 5 being of diagnostic quality.
Lesion Detectability | through study completion, an average of 1 year
  Three (3) qualified Nuclear Medicine Physicians shall complete a lesion detectability evaluation of the SoC PET/CT scan (as determined in Phase 1) and OMNI PET/CT scan for each lesion identified for each subject.
  Each reader will evaluate the reconstructed images by qualitatively evaluating the visibility of the lesions and by measuring the relevant quantitative values of glycolytic activity of each suspicious lesion (contrast, noise, SUV). The variables conventionally used to quantify the glycolytic activity in PET for characterization, prognosis and therapeutic monitoring are as follows:
  * SUV (Standardized Uptake Value): SUVmax, SUVmean, SUVpeak
  * Metabolically active volume: VMA
  * Total glycolysis of the lesion: TLG = SUV x VMA The reader shall provide the location information of each identified lesion.

CONTACTS AND LOCATIONS:
Overall Officials: Brian W Thomsen, Study Director — GE Healthcare
Locations (1):
- Institut Claudius Regaud, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Maronnier Q, Cassou-Mounat T, Gabiache E, Latge A, Terroir M, Vija L, Su KH, Caselles O, Courbon F. Deep learning-enhanced digital-BGO versus TOF PET/CT: comparative assessment of detection, quantitation, and overall image quality. EJNMMI Phys. 2025 Dec 16. doi: 10.1186/s40658-025-00814-8. Online ahead of print. PMID 41400899